CLINICAL TRIAL: NCT01037738
Title: Intraarticular Application of Autologous Conditioned Serum (ACS/Orthokine) Reduces Bone Tunnel Widening After ACL Reconstructive Surgery A Prospective, Randomized, Saline-controlled, Patient- and Observer-blinded, Parallel-design Trial
Brief Title: Study of Autologous Conditioned Serum After Anterior Cruciate Ligament Reconstructive Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Zagreb (Other)
Collaborators: Croatian Institute of Health Insurance (Unknown)
Responsible Party: Nikica Darabos, MD PhD, University Clinic for Traumatology, Draskoviceva 19, 10000 Zagreb, Croatia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REC LCA 2B
Record Dates: First submitted 2009-12-03; First posted 2009-12-23 (Estimated); Last update posted 2009-12-23 (Estimated); Status verified 2009-01

CONDITIONS: Joint Instability
Keywords: ACL reconstruction; autologous conditioned serum; Orthokine; osteoarthritis; interleukin receptor antagonist; growth factors; WOMAC; IKDC
MeSH Terms: conditions — Joint Instability; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ACS - Orthokin (Active Comparator): Autologous conditioned serum (ACS) - Orthokin containing endogenous anti-inflammatory cytokines including IL-1Ra and growth factors (IGF-1, PDGF and TGF-ß1, among others) in the liquid blood phase.
  Interventions: Procedure: ACL reconstructive surgery and ACS/ Orthokin application
- Placebo (Placebo Comparator): Physiologic solution
  Interventions: Procedure: ACL reconstructive surgery and ACS/ Orthokin application

INTERVENTIONS:
Procedure: ACL reconstructive surgery and ACS/ Orthokin application — ACL reconstructive surgery and ACS/ Orthokin or Placebo intraarticular application on Day 0,1,6 and 10 postoperatively, regarding the Arm

SUMMARY:
Abstract

Background

Pro-inflammatory cytokines play a pivotal role in osteoarthritis, as well as in bone tunnel widening after ACL reconstructive surgery. A new treatment option is to administer autologous conditioned serum (ACS) containing endogenous anti-inflammatory cytokines including IL-1Ra and growth factors (IGF-1, PDGF and TGF-ß1, among others) in the liquid blood phase.

Objective The purpose of this trial was to establish whether the osteoclastic effect could be affected by intra-articular application of ACS, thus resulting in a potential decrease of knee laxity and leading to a better postoperative outcome.

Methods In a prospective, randomized, double-blinded, placebo-controlled trial with two parallel groups, 62 patients were treated. Bone tunnel width was measured by CT scans, while clinical efficacy was assessed by patient-administered outcome instruments (WOMAC, IKDC 2000) up to one year following the ACL reconstruction in patients receiving either ACS (Group A) or placebo (Group B). The investigators compared the levels and dynamics of IL-1b concentrations in the synovial liquid and examined the correlation between the levels of IL-1b at three different post-operative points.

Level of evidence Therapeutic study, Level 1 (randomized controlled trial [significant differences and narrow confidence intervals])

ELIGIBILITY:
Inclusion Criteria:

Eligible patients were:

* older than 18 years
* prior to each surgery, traumatic ACL rupture was determined on the basis of a clinical examination and confirmed by exploratory and therapeutic arthroscopic surgery in accordance with good surgical practice
* the same preoperative diagnosis of isolated ACL rupture
* a knee axis deviation up to 5°; knee osteoarthritis up to grade 1 according to the AO
* knee chondral lesion up to grade 2 (Outerbridge classification).

Exclusion Criteria:

* poor general health as judged by the orthopedic surgeon
* Concomitant painful or disabling disease of the spine, hips, or lower limbs that would interfere with evaluation of the afflicted knee
* Any clinically significant or symptomatic vascular or neurological disorder; crystalline, inflammatory and infectious arthropathies
* Infections
* Osteomyelitis
* Alcohol/drug abuse
* Known coagulopathy
* Corticosteroid or anti-coagulant usage, and morbid obesity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2006-05; Primary Completion 2008-08 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Bone tunnel width - CT scans. Clinical efficacy - patient administered outcome instruments (WOMAC, IKDC 2000). | 1 year

SECONDARY OUTCOMES:
Measurements and correlation between the levels of synovial fluid IL-1b at three different post-operative points. | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Medical School, University of Zagreb, Zagreb, Croatia

REFERENCES:
- [Background] References 1. Harris NL, Indelicato PA, Bloomberg MS, Meister K, Wheeler DL. Radiographic and histologic analysis of the tibial tunnel after allograft anterior cruciate ligament reconstruction in goats. American Journal of Sports Medicine 30 (3):368-73,2002. 2. Hoher J, Moller HD, Fu FH. Bone tunnel enlargement after anterior cruciate ligament reconstruction: fact or fiction? Knee Surgery, Sports Traumatology and Arthroscopy 6 (4):231-40,1998. 3. Hsu CJ, Hsu HC, Jim YF. A radiological study after anterior cruciate ligament reconstruction. Journal of Chinese Medical Association 66(3):160-5,2003. 4. Nakayama Y, Shirai Y, Narita T, Mori A. Enlargement of bone tunnels after anterior cruciate ligament reconstruction. Nippon Ika Daigaku Zasshi 65(5):377-81,1998. 5. Topliss C, Webb J. An audit of tunnel position in anterior cruciate ligament reconstruction. Knee 8(1):59-63,2001.